CLINICAL TRIAL: NCT02792855
Title: Randomized Study Comparing the "snifﬁng Position" , "Simple Head Extension" and "Neutral Position" for Awake Orotracheal Intubation With Fiberoptic in Anticipate Difficult Airway Patients
Brief Title: Comparing the "snifﬁng Position" , "Simple Head Extension" and "Neutral Position"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 9958
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2020-11

CONDITIONS: Therapeutic Procedural Complication
Keywords: Snifﬁng Position; Simple Head Extension; neutral position

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- snifﬁng Position (Experimental): Awake fiberoptic bronchoscope(FOB) orotracheal under snifﬁng position.The snifﬁng position was obtained by placement of a 7-cm cushion under the head of the patient. When the FOB was inserted into oral cavity, and the epiglottis and glottis were identified by the FOB. The anterior of FOB was inserted deep into tracheal after the glottis was exposed sufficiently then the tracheal tube was pushed into the trachea via the FOB
  Interventions: Device: snifﬁng Position(place a 7-cm cushion under head )
- Simple Head Extension (Experimental): Awake fiberoptic bronchoscope(FOB) orotracheal under Head Extension position.The Head Extension position was obtained by simple head extension.When the FOB was inserted into oral cavity, and the epiglottis and glottis were identified by the FOB. The anterior of FOB was inserted deep into tracheal after the glottis was exposed sufficiently then the tracheal tube was pushed into the trachea via the FOB
  Interventions: Device: Simple Head Extension(without cushion)

INTERVENTIONS:
Device: snifﬁng Position(place a 7-cm cushion under head ) — Awake fiberoptic bronchoscope(FOB) orotracheal under snifﬁng position.The snifﬁng position was obtained by placement of a 7-cm cushion under the head of the patient. When the FOB was inserted into oral cavity, and the epiglottis and glottis were identified by the FOB. The anterior of FOB was inserted deep into tracheal after the glottis was exposed sufficiently then the tracheal tube was pushed into the trachea via the FOB
  Arms: snifﬁng Position
Device: Simple Head Extension(without cushion) — Awake fiberoptic bronchoscope(FOB) orotracheal under Head Extension position.The Head Extension position was obtained by simple head extension.When the FOB was inserted into oral cavity, and the epiglottis and glottis were identified by the FOB. The anterior of FOB was inserted deep into tracheal after the glottis was exposed sufficiently then the tracheal tube was pushed into the trachea via the FOB
  Arms: Simple Head Extension

SUMMARY:
The simple head extension is recommended for optimization of glottic visualization during awake orotracheal intubation whith fiberoptic bronchoscope (FOB) . However, no study to date has conﬁrmed its superiority over "snifﬁng position" . In a prospective, randomized study, the authors compared the snifﬁng position , simple head extension and "Neutral Position" in awake orotracheal Intubation.

DETAILED DESCRIPTION:
The study included seventy-five patients with anticipated difficult airways. The snifﬁng position was obtained by placement of a 7-cm cushion under the head of the patient. The extension head position was obtained by by placement of a 7-cm cushion under the shoulder.

The head position was randomized as follows: neutral position group (NP group), sniffing position group (SP group) or extension position group (EP group) Randomization was performed by placing index cards with the letter NP or SP or EP into75 sealed envelopes , which were then placed in random order. At the time of a patient's enrollment, the next available envelope was placed with the patient's chart. At the time of intubation, the envelope was opened and the sequence was thus determined.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than 30 kg/m2
* ASA classifications of I-II, modified Mallampati classification of 3 or 4, requiring general anesthesia were included.

Exclusion Criteria:

* Exclusion criteria included age younger than 18 yr
* ASA class IV or V
* Abnormalities of the heart, brain, liver, lung, kidney and coagulation functions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Intubation Time | Ten minutes
  The primary endpoints were the time to view the vocal cords (TVC) which was taken when the operator indicated verbally that he view the vocal cords and the time to successful tracheal intubation (TSI). TSI was defined as the time taken from insertion of the FOB between the teeth until the appearance of a capnograhy curve.

SECONDARY OUTCOMES:
Occurrence of throat pain measured by VAS | one day Postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ximing Qi, Study Director — The First Hospital of Qinhuangdao
Locations (1):
- 中国, Qinhuangdao, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Liu Z, Zhao L, Ma Z, Liu M, Qi X, Jia Q, Liang S, Yang X. Effects of head positions on awake fiberoptic bronchoscope oral intubation: a randomized controlled trial. BMC Anesthesiol. 2021 Jun 23;21(1):176. doi: 10.1186/s12871-021-01397-4. PMID 34162330